CLINICAL TRIAL: NCT03124082
Title: Study Protocol "OFA: Opioid-Free Anesthesia".
Brief Title: OFA - Opioid Free Anesthesia
Acronym: OFA
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Parma (Other)
Responsible Party: Principal Investigator, Massimo Allegri, MD, Assistant Professor, University of Parma
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 34477
Record Dates: First submitted 2017-01-22; First posted 2017-04-21 (Actual); Last update posted 2017-04-21 (Actual); Status verified 2017-04

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Remifentanil; Ketamine; Lidocaine; Clonidine

STUDY DESIGN:
Intervention Model Description: randomized double blind trial
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- opioid (Active Comparator): remifentanil 0,15-0,25 mcg/kg/h
  Interventions: Drug: Remifentanil
- opioid free (Experimental): ketamine bolus 0,5 mg/kg + infusion 0,25 mg/kg/h lidocaine bolus 1 mg/kg + infusion 1 mg/kg/h clonidine 4 mcg/kg
  Interventions: Drug: Ketamine; Drug: Lidocaine; Drug: Clonidine

INTERVENTIONS:
Drug: Remifentanil — continuous infusion intraop
  Arms: opioid
Drug: Ketamine — bolus 0,5 mg/kg + infusion 0,25 mg/kg/h
  Arms: opioid free
Drug: Lidocaine — lidocaine bolus 1 mg/kg + infusion 1 mg/kg/h
  Arms: opioid free
Drug: Clonidine — clonidine 4 mcg/kg
  Arms: opioid free

SUMMARY:
Opioids have been used for analgesia since many years, but despite potent analgesia they are also associated to side effects, including opioid induced Hyperalgesia (OIH).

OIH in the surgical setting is debated, and may predispose patients to higher analgesic consumption in the preoperative period, and peripheral and central sensitization. The aim of the study is to compare remifentanil-based vs non opioid analgesia (clonidine, lidocaine, ketamine) for intraoperative management of patients undergoing laparoscopic left hemicolectomy, with the hypothesis that non- opiod treated patients will have lower morphine consumption in the first 24 hours after surgery. Peripheral and central hyperalgesia will be tested with Von Frey hairs and pin-prick to evaluate acute CNS (Central Nervous System) sensitization after surgery. Acute and persistent (1 and 3 months) pain will be registered, together with any side effect and parameters of surgical rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* left hemicolectomy
* signed informed consent
* >18 ys

Exclusion Criteria:

* >90 ys <18 ys
* no consent
* pregnancy
* psychiatric disease
* cardiac failure, aortic or mitral valve severe stenosis
* kidney or hepatic failure
* atrio-ventricular type II block
* immunodepression
* emergency surgery
* ICU admittance
* drug or alcohol abuse
* chronic pain

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2017-01-04 (Actual); Primary Completion 2017-12-31 (Estimated); Study Completion 2018-03-31 (Estimated)

PRIMARY OUTCOMES:
analgesic consumption | 24 HOURS
  morphine mg by PCA (Patient Controlled Analgesia)

SECONDARY OUTCOMES:
side effects | 4 days after surgery
  nausea and vomiting, ileus, itching, shiver, hypotension, bradycardia, sedation
Pain Score on the Visual Analog Scale | 3 months
  VAS (Visual Analog Scale)
peripheral sensitization | 24 hours
  assessment of primary hyperalgesia by Von Frey Filaments at 24 hours
central sensitization | 24 hours
  assessment of secondary hyperalgesia by pin-prick test at 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Parma, Parma, Italy

IPD SHARING:
Plan to Share IPD: No